CLINICAL TRIAL: NCT00516893
Title: A Multicenter, Open-Label Immunogenicity and Safety Study of Natalizumab High Titer Material (BG00002-E) in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: Natalizumab High Titer Immunogenicity and Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Biogen Idec Medical Director, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 101MS201
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis
Keywords: natalizumab; Tysabri; Multiple Sclerosis; Relapsing Forms of Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab High Titer (Experimental): natalizumab high titer 300 mg administered as intravenous (IV) infusion over 60 minutes once every 4 weeks for up to 9 doses
  Interventions: Biological: BG00002-E (natalizumab high titer)

INTERVENTIONS:
Biological: BG00002-E (natalizumab high titer)
  Other Names: Tysabri

SUMMARY:
The primary objective of the study was to evaluate the immunogenicity of natalizumab (Tysabri®) produced by a modified manufacturing process (natalizumab high titer; BG00002-E) administered intravenously (IV) to participants with relapsing forms of multiple sclerosis (MS). The secondary objective of this study was to evaluate the safety of natalizumab high titer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a relapsing form of MS
* Must fall within the therapeutic indications stated in the locally approved label for natalizumab
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Prior treatment with natalizumab
* Considered by investigator to be immunocompromised
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (13):
- United States (13):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Farmington Hills, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research site, Round Rock, Texas
  - Research Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natalizumab High Titer
Started | 113
Received Study Treatment | 112
Completed | 92
Not Completed | 21
Not completed — Lost to Follow-up | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Noncompliance | 2
Not completed — Death | 1
Not completed — Persistent Antibodies per Protocol | 6
Not completed — Relocated | 1
Not completed — Pregnancy | 1
Not completed — Received Medication From Another Study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Natalizumab High Titer
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.64)
Age, Customized [Number; unit: participants] — Protocol deviations were filed for the 2 participants >=56 years.
  participants
    ≥ 18 to < 20 years | 2
    ≥ 20 to < 30 years | 15
    ≥ 30 to < 40 years | 43
    ≥ 40 to < 50 years | 41
    ≥ 50 to < 56 years | 10
    ≥ 56 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 8
  Asian | 1
  White | 91
  Hispanic | 12
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 113
Expanded Disability Status Score (EDSS) Score [Mean (Standard Deviation); unit: scores on a scale] — EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. All participants who were dosed (n=112) had an EDSS baseline score recorded.
  scores on a scale | 3.66 (1.817)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-Natalizumab Antibody Negative, Transient Positive, and Persistent Positive Status
Description: Negative: no detectable antibody at all post-baseline visits. Persistent positive: antibody positive at 2 or more post-baseline visits at least 42 days apart, or positive at the last post-baseline visit. Transient positive: antibody positive at only 1 post-baseline visit prior to the last visit.
Time Frame: Assessed every 12 weeks from Week 0 (Baseline) to Week 36
Population: Participants who received at least 1 dose of natalizumab, had a negative baseline antibody result, and had at least 1 antibody assessment after the first dose.
Measure: Number; unit: participants
Arm/Group | Natalizumab High Titer
Number analyzed (Participants) | 108
participants
  Antibody negative | 96
  Transient positive | 3
  Persistent positive | 9

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: AE: any sign, symptom, or diagnosis/disease that was unfavorable or unintended, new, or if pre-existing, worsened in a participant administered a study treatment and that did not necessarily have a causal relationship with this treatment. SAE: an event that resulted in death; an event that, in the view of the investigator, placed the participant at immediate risk of death (life-threatening event); an outcome that resulted in a congenital anomaly/birth defect diagnosed in a child of a participant in this study; an event that required or prolonged inpatient hospitalization; an event that resulted in persistent or significant disability/incapacity; any other medically important event that, in the opinion of the investigator, may have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed above. Events were classified as 'related' or 'not related' to study drug, and categorized as 'mild' moderate' or 'severe' per protocol.
Time Frame: AEs: collected from Baseline (Week 0) until Week 36 or premature withdrawal. SAEs: collected from informed consent until Week 36 or premature withdrawal.
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Natalizumab High Titer
Number analyzed (Participants) | 112
participants
  Adverse event (AE) | 106
  Moderate or severe AE | 63
  Severe AE | 18
  AE related to study drug | 23
  Serious adverse event (SAE) | 7
  SAE related to study drug | 0
  Treatment discontinuation due to AE | 4
  Withdrawal from study due to AE | 3

3. Secondary Outcome: Mean Change From Baseline in Expanded Disability Status Scale (EDSS) Scores at Week 36
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. The change in EDSS at Month 36 was calculated as EDSS at Month 36 minus EDSS at baseline.
Time Frame: Baseline, Week 36
Population: Participants with EDSS scores at Baseline and Week 36 (includes participants who withdrew from the study).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Natalizumab High Titer
Number analyzed (Participants) | 106
scores on a scale | -0.19 (0.982)

4. Secondary Outcome: Annualized Relapse Rate
Description: Annualized relapse rate was calculated as the total number of relapses that occurred during the study divided by the total number of years the participant was followed in the study. The annualized relapse rate was based only on those relapses that were determined to meet the definition of relapse per the investigator's clinical judgment. New or recurrent symptoms that occurred less than 30 days following the onset of a protocol-defined relapse were considered part of the same relapse.
Time Frame: Through Week 36
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: relapses/participant-years
Arm/Group | Natalizumab High Titer
Number analyzed (Participants) | 112
relapses/participant-years | 0.13

ADVERSE EVENTS:
Time Frame: AEs: collected from Baseline (Week 0) until Week 36 or premature withdrawal. SAEs: collected from informed consent until Week 36 or premature withdrawal.
Description: Includes all participants who received at least 1 dose of study drug.
Arm/Group | Natalizumab High Titer
Serious Adverse Events (participants affected / at risk) | 7/112
Other Adverse Events (participants affected / at risk) | 79/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab High Titer (N=112)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Multiple sclerosis relapse (Nervous system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (Vascular disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Demyelination (Nervous system disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab High Titer (N=112)
Headache (Nervous system disorders) | 22
Fatigue (General disorders) | 20
Upper respiratory tract infection (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 12
Sinusitis (Infections and infestations) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Fall (Injury, poisoning and procedural complications) | 10
Multiple sclerosis relapse (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7
Contusion (Injury, poisoning and procedural complications) | 7
Visual acuity reduced (Eye disorders) | 7
Gait disturbance (General disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Nasopharyngitis (Infections and infestations) | 6
Vision blurred (Eye disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.